CLINICAL TRIAL: NCT05481879
Title: A Randomized, Placebo-Controlled, Multiple Ascending Dose Study Assessing Safety, Tolerability, Pharmacodynamics, Efficacy, and Pharmacokinetics of DYNE-101 Administered to Participants With Myotonic Dystrophy Type 1
Brief Title: Safety, Tolerability, Pharmacodynamic, Efficacy, and Pharmacokinetic Study of DYNE-101 in Participants With Myotonic Dystrophy Type 1
Acronym: ACHIEVE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dyne Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DYNE101-DM1-201; 2023-510353-42-00 (EU CTIS Number)
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-08

CONDITIONS: Myotonic Dystrophy Type 1 (DM1)
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- MAD Cohort: Placebo-Controlled Period: DYNE-101 (Experimental): Participants will be randomized to receive ascending doses of DYNE-101, once every 4 weeks (Q4W) or once every 8 weeks (Q8W) for up to 24 weeks.
  Interventions: Drug: DYNE-101
- MAD Cohort: Placebo-Controlled Period: Placebo (Placebo Comparator): Participants will be randomized to receive DYNE-101 matching placebo, Q4W or Q8W for up to 24 weeks.
  Interventions: Drug: Placebo
- MAD Cohort: Treatment Period: DYNE-101 (Experimental): Participants who receive DYNE-101 in Placebo-Controlled Period will continue to receive DYNE-101, Q4W or Q8W for up to 24 weeks.
  Participants who receive placebo in Placebo-Controlled Period will receive DYNE-101, Q4W or Q8W for up to 24 weeks.
  Interventions: Drug: DYNE-101; Drug: Placebo
- MAD Cohort: Long-Term Extension Period: DYNE-101 (Experimental): Participants will receive DYNE-101, Q4W or Q8W for up to 168 weeks.
  Interventions: Drug: DYNE-101
- Dose Expansion Cohort: Placebo-Controlled Period: DYNE-101 (Experimental): Participants will receive DYNE-101, Q8W for up to 24 weeks.
  Interventions: Drug: DYNE-101
- Dose Expansion Cohort: Placebo-Controlled Period: Placebo (Experimental): Participants will receive DYNE-101 matching placebo, Q8W for up to 24 weeks.
  Interventions: Drug: Placebo
- Dose Expansion Cohort: Treatment Period: DYNE-101 (Experimental): Participants who receive DYNE-101 in Placebo-Controlled Period will continue to receive DYNE-101, Q8W for up to 24 weeks.
  Participants who receive placebo in Placebo-Controlled Period will receive DYNE-101, Q8W for up to 24 weeks.
  Interventions: Drug: DYNE-101; Drug: Placebo
- Dose Expansion Cohort: Long-Term Extension Period: DYNE-101 (Experimental): Participants will receive DYNE-101, Q8W for up to 168 weeks.
  Interventions: Drug: DYNE-101

INTERVENTIONS:
Drug: DYNE-101 — Administered by IV infusion
  Arms: Dose Expansion Cohort: Long-Term Extension Period: DYNE-101; Dose Expansion Cohort: Placebo-Controlled Period: DYNE-101; Dose Expansion Cohort: Treatment Period: DYNE-101; MAD Cohort: Long-Term Extension Period: DYNE-101; MAD Cohort: Placebo-Controlled Period: DYNE-101; MAD Cohort: Treatment Period: DYNE-101
Drug: Placebo — Administered by IV infusion
  Arms: Dose Expansion Cohort: Placebo-Controlled Period: Placebo; Dose Expansion Cohort: Treatment Period: DYNE-101; MAD Cohort: Placebo-Controlled Period: Placebo; MAD Cohort: Treatment Period: DYNE-101

SUMMARY:
The primary purpose of the study is to evaluate the safety and tolerability of multiple intravenous (IV) doses of DYNE-101 administered to participants with Myotonic Dystrophy Type 1 (DM1).

The study consists of 4 periods: A Screening Period (up to 8 weeks), a Placebo-Controlled Period (24 weeks), a Treatment Period (24 weeks) and a Long-Term Extension (LTE) Period (168 weeks) in both multiple-ascending dose (MAD) and dose expansion cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DM1 with trinucleotide repeat size >100.
* Age of onset of DM1 muscle symptoms ≥12 years.
* Clinically apparent myotonia equivalent to hand opening time of at least 2 seconds in the opinion of the Investigator.
* Hand grip strength and ankle dorsiflexion strength.
* Able to complete 10-MWRT, stair ascend/descend (MAD cohorts only), and 5×STS at screening without the use of assistive devices such as canes, walkers, or orthoses.

Exclusion Criteria:

* History of major surgical procedure within 12 weeks prior to the start of investigative product administration or an expectation of a major surgical procedure (eg, implantation of cardiac defibrillator) during the study.
* History of anaphylaxis.
* Medical condition other than DM1 that would significantly impact ambulation or participation in functional assessments.
* Treatment with medications that can improve myotonia within a period of 5 half-lives of the medication prior to performing screening assessments.
* Electrocardiogram (ECG) with the corrected QT interval by Fridericia's Formula (QTcF) ≥450 milliseconds (ms) in men and QTcF ≥460 ms in women, PR ≥240 ms, left bundle-branch block, or a conduction defect, which is clinically significant in the opinion of the Investigator.
* Percent predicted forced vital capacity (FVC) <50%.
* History of tibialis anterior biopsy within 3 months of Day 1 or planning to undergo tibialis anterior biopsies during study period for reasons unrelated to the study.
* Participant has a history of suicide attempt, suicidal behavior, or has any suicidal ideation within 6 months prior to Screening that meets criteria at a level of 4 or 5 of the Columbia Suicide Severity Rating Scale (C-SSRS) or who, in the opinion of the Investigator, is at significant risk to commit suicide.
* Use of glucagon-like peptide 1 (GLP-1) agonist medications including semaglutide, dulaglutide, liraglutide, exenatide, or tirzepatide within a period of 5 half-lives of the medication prior to performing screening assessments.
* Significant weight loss during study participation may impact weight-based dosing, performance on muscle function assessments, and pharmacodynamic (PD) biomarkers.

Note: Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
MAD Cohorts: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | Through study completion, up to Week 217
Dose Expansion Cohorts: Change From Baseline in Myotonia as Measured by Video Hand Opening Time (vHOT) | Baseline up to Week 25

SECONDARY OUTCOMES:
MAD Cohorts: Change From Baseline in Composite Alternative Splicing Index (CASI) in Skeletal Muscle Tissue | Baseline up to Week 45
MAD Cohorts: Change From Baseline in Dystrophia Myotonica Protein Kinase (DMPK) Ribonucleic Acid (RNA) Expression in Muscle Tissue | Baseline up to Week 45
MAD Cohorts: Change From Baseline in Hand Grip Relaxation Time | Baseline up to Week 121
MAD Cohorts: Change From Baseline in Myotonia as Measured by vHOT | Baseline up to Week 193
MAD Cohorts: Change From Baseline in Quantitative Myometry Testing (QMT) | Baseline up to Week 193
MAD Cohorts: Change From Baseline in 10-Meter Walk/Run Test (10-MWRT) | Baseline up to Week 193
MAD Cohorts: Change From Baseline in Stair-Ascend/Descend Test | Baseline up to Week 121
MAD Cohorts: Change From Baseline in 5 Times Sit to Stand (5×STS) | Baseline up to Week 193
MAD Cohorts: Change From Baseline in 9-Hole Peg Test (9-HPT) | Baseline up to Week 193
MAD Cohorts: Maximum Observed Plasma Drug Concentration (Cmax) of DYNE-101 | Pre-dose, and at multiple timepoints up to Week 217
MAD Cohorts: Time to Maximum Observed Plasma Concentration (tmax) of DYNE-101 | Pre-dose, and at multiple timepoints up to Week 217
MAD Cohorts: Area Under the Concentration-time Curve From Hour 0 to the Last Measurable Plasma Concentration (AUCtlast) of DYNE-101 | Pre-dose, and at multiple timepoints up to Week 217
MAD Cohorts: Area Under the Concentration-time Curve Extrapolated to Infinity (AUC∞) of DYNE-101 in Plasma | Pre-dose, and at multiple timepoints up to Week 217
MAD Cohorts: Apparent Terminal Elimination Rate Constant (λz) of DYNE-101 in Plasma | Pre-dose, and at multiple timepoints up to Week 217
MAD Cohorts: Apparent Terminal Elimination Half-Life (t1/2) of DYNE-101 in Plasma | Pre-dose, and at multiple timepoints up to Week 217
MAD Cohorts: Clearance (CL) of DYNE-101 in Plasma | Pre-dose, and at multiple timepoints up to Week 217
MAD Cohorts: Volume of Distribution at the Terminal Phase (Vz) of DYNE-101 in Plasma | Pre-dose, and at multiple timepoints up to Week 217
MAD Cohorts: Volume of Distribution at Steady State (Vss) of DYNE-101 in Plasma | Pre-dose, and at multiple timepoints up to Week 217
MAD Cohorts: Antisense Oligonucleotide (ASO) Concentration of DYNE-101 in Muscle Tissue | Up to Week 45
MAD Cohorts: Number of Participants With Antidrug Antibodies (ADAs) | Up to Week 217
Dose Expansion Cohorts: Change From Baseline in CASI in Skeletal Muscle Tissue | Baseline up to Week 25
Dose Expansion Cohorts: Change From Baseline in QMT Total | Baseline up to Week 25
Dose Expansion Cohorts: Change From Baseline in 10-MWRT | Baseline up to Week 25
Dose Expansion Cohorts: Change From Baseline in 5×STS | Baseline up to Week 25
Dose Expansion Cohorts: Change From Baseline in 9-HPT | Baseline up to Week 25
Dose Expansion Cohorts: Change From Baseline in Myotonic Dystrophy Health Index (MDHI) Total Score | Baseline up to Week 25
Dose Expansion Cohorts: Patient Global Impression of Change (PGI-C) | Baseline up to Week 25
Clinician Global Impression of Change (CGI-C) | Baseline up to Week 25
Dose Expansion Cohorts: Change From Baseline in Patient Global Impression of Severity (PGI-S) | Baseline up to Week 25
Dose Expansion Cohorts: Change From Baseline in Clinician Global Impression of Severity (CGI-S) | Baseline up to Week 25
Dose Expansion Cohorts: Change From Baseline in MDHI Subscale Scores | Baseline up to Week 25
Dose Expansion Cohorts: Change From Baseline at in Myotonic Dystrophy type 1 Activity and Participation Scale (DM1-ACTIV^C) Total Score | Baseline up to Week 25
Dose Expansion Cohorts: Change From Baseline in Percent Predicted Hand Grip Strength | Baseline up to Week 25

CONTACTS AND LOCATIONS:
Locations (16):
- United States (5):
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Rochester Medical Center, Rochester, New York
  - Neurology Rare Disease Center, Denton, Texas
  - Virginia Commonwealth University (VCU), Richmond, Virginia
- St. Vincent's Hospital, Fitzroy, Victoria, Australia
- France (2):
  - CHU de Nantes, Nantes
  - Institut de Myologie, Paris
- Ludwig Maximilians University, Munich - Friedrich Baur Institut, Munich, Germany
- Italy (2):
  - Centro Clinico Nemo, Milan
  - Fondazione Policlinico Universitario A Gemelli-Rome, Rome
- Radboud Medical Center, Nijmegen, Netherlands
- NZCR Auckland, Auckland, New Zealand
- United Kingdom (3):
  - University College London Hospitals, London
  - John Walton Muscular Dystrophy Research Centre, Newcastle upon Tyne
  - Salford Royal Hospital, Salford

IPD SHARING:
Plan to Share IPD: No